CLINICAL TRIAL: NCT02998905
Title: Non-Vitamin K Antagonist Oral Anticoagulants for Stroke Prevention in Patients With Atrial Fibrillation and Previous Intracerebral Hemorrhage Study
Brief Title: NOACs for Stroke Prevention in Patients With Atrial Fibrillation and Previous ICH
Acronym: NASPAF-ICH
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Population Health Research Institute (Other)
Responsible Party: Principal Investigator, Ashkan Shoamanesh, Assistant Professor of Medicine (Neurology), Population Health Research Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NASPAF-ICH
Record Dates: First submitted 2016-11-25; First posted 2016-12-21 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Atrial Fibrillation; Intracerebral Hemorrhage
MeSH Terms: conditions — Atrial Fibrillation; Cerebral Hemorrhage | interventions — N(4)-oleylcytosine arabinoside; Aspirin

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NOAC (Experimental): Apixaban or dabigatran or edoxaban or rivaroxaban
  Interventions: Drug: NOAC
- Acetylsalicylic Acid (Active Comparator): Acetylsalicylic acid
  Interventions: Drug: Acetylsalicylic Acid

INTERVENTIONS:
Drug: NOAC — Apixaban or dabigatran or edoxaban or rivaroxaban at recommended dosing for stroke prevention in atrial fibrillation. The particular agent is at the discretion of the local investigator.
  Arms: NOAC
Drug: Acetylsalicylic Acid — Acetylsalicylic acid 81 mg/day
  Arms: Acetylsalicylic Acid

SUMMARY:
To determine the feasibility of a controlled trial examining the efficacy and safety of non-vitamin K antagonist oral anticoagulants (NOACs) compared with ASA for stroke prevention in patients with a high-risk of atrial fibrillation and previous intracerebral hemorrhage.

DETAILED DESCRIPTION:
The NASPAF-ICH study is an open-label, randomized, controlled, phase II study that will assess the feasibility of a controlled trial examining the efficacy and safety of non-vitamin K antagonist oral anticoagulants (NOACs) compared with acetylsalicylic acid (ASA) for stroke prevention in patients with high-risk atrial fibrillation and previous intracerebral hemorrhage, as well as provide evidence of efficacy and safety for planning of a phase III trial. Recruitment will occur at 10 high-volume stroke research centres across Canada over 2 years, at which 100 adult patients with high-risk atrial fibrillation (CHADS2 ≥2) and previous spontaneous or traumatic ICH (intraparenchymal or intraventricular hemorrhage while on or off anticoagulation) will be randomly assigned to receive a NOAC (particular agent at the discretion of the local investigator) or ASA 81 mg per day. Patients will be followed for a mean of 1 year to a common end-study date. The feasibility of recruitment will also be tested. The investigators estimate that five patients per year per centre can be recruited.

ELIGIBILITY:
Inclusion Criteria:

* Previous primary intracerebral hemorrhage
* Atrial fibrillation (CHADS2 ≥ 2)

Exclusion Criteria:

* Non-stroke indication for antiplatelet or anticoagulant therapy
* Recent intracerebral hemorrhage within 14 days
* Platelet count less than 100,000/mm3 at enrollment or other bleeding diathesis
* Prior symptomatic lobar intracerebral hemorrhage other than the qualifying event
* Uncontrollable hypertension consistently above SBP/DBP of 160/100 mmHg
* Known hypersensitivity to either ASA or NOACs
* Inability to adhere to study procedures

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-26 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2020-02-18 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | Through study completion; ~ 30 months
  The mean number of patients randomized per site per year.
Composite of ischemic stroke and recurrent intracerebral hemorrhage | Through study completion; average of 1 year
  The composite of ischemic stroke and recurrent intracerebral hemorrhage

SECONDARY OUTCOMES:
Refusal rate | Through study completion; average of 1 year
  Average number of eligible patients per site who refuse consent.
Retention rate | Through study completion; average of 1 year
  Randomized patients who completed 6 months of follow-up on drug or died during trial participation.
Ischemic stroke | Through study completion; average of 1 year
  Development of an acute neurologic deficit in conjunction with brain imaging consistent with acute/subacute ischemic stroke.
Intracerebral hemorrhage | Through study completion; average of 1 year
  A neurologic deficit associated with an intraparenchymal or intraventricular hemorrhage on computed tomography (CT) or MRI scan, or as demonstrated by surgery or autopsy.
Fatal stroke | Through study completion; average of 1 year
  Death that is attributable to an ischemic stroke or intracerebral hemorrhage.
Myocardial infarction | Through study completion; average of 1 year
  Defined by presence of at least one of the following a compatible clinical history and characteristic serum enzymes changes with or without electrocardiographic abnormalities; clinical history and serial ST-segment and T-wave changes which are specifically located with respect to the electrocardiographic leads accompanied by elevation of CPK-MB isoenzyme or troponin in serum; the development of large Q-waves on electrocardiography associated with changes in the ST-segments and T-waves in specific and appropriate leads which indicate the location of the infarct, even in the absence of symptoms or abnormalities in serum enzymes; development of discrete, segmental left ventricular systolic wall motion abnormality concurrent with compatible clinical history, electrocardiographic changes or serum enzyme abnormalities; or histopathological evidence of subacute myocardial necrosis.
All-cause mortality | Through study completion; average of 1 year
  Persistent and irreversible absence of brain or brainstem function.
Systemic thromboembolism | Through study completion; average of 1 year
  Emboli to the arterial circulation excluding myocardial infarction, ischemic stroke or intracerebral hemorrhage.
Major hemorrhage | Through study completion; average of 1 year
  Bleeding accompanied by one or more of the following - a decrease in the hemoglobin level of ≥20 g per liter over a 24-hour period, transfusion of ≥2 units of packed red cells, bleeding at a critical site (intracranial, intraspinal, intraocular, pericardial, intraarticular, intramuscular with compartment syndrome, or retroperitoneal), or fatal bleeding.
Intracranial hemorrhage | Through study completion; average of 1 year
  Signs or symptoms associated with an epidural, subdural, subarachnoid, intraparenchymal or intraventricular hemorrhage on computed tomography (CT) or MRI scan, or as demonstrated by surgery or autopsy.
Composite of all stroke, myocardial infarct, systemic thromboembolism or death | Through study completion; average of 1 year
  Composite of all stroke, myocardial infarct, systemic thromboembolism or death
Modified Rankin Scale (mRS) | Through study completion; average of 1 year
  Average mRS score
Montreal Cognitive Assessment (MOCA) | Through study completion; average of 1 year
  Average MOCA score

OTHER OUTCOMES:
Weighted net clinical benefit | Through study completion; average of 1 year
  Weighted net clinical benefit factoring the impact of ischemic stroke, intracerebral hemorrhage, non-intracerebral intracranial hemorrhage, major extracranial hemorrhage and myocardial infarction on death and disability.

CONTACTS AND LOCATIONS:
Overall Officials: Ashkan Shoamanesh, MD FRCPC, Principal Investigator — Population Health Research Institute
Locations (9):
- Canada (9):
  - Foothills Medical Centre, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Vancouver Coastal Health Research Institute, Vancouver, British Columbia
  - Hamilton Health Sciences, Hamilton, Ontario
  - London Health Sciences Centre - University Hospital, London, Ontario
  - The Ottawa Hospital Research Institute, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Toronto Western Hospital, Toronto, Ontario
  - Hopital Notre-Dame du CHUM, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cochrane A, Chen C, Stephen J, Ronning OM, Anderson CS, Hankey GJ, Al-Shahi Salman R. Antithrombotic treatment after stroke due to intracerebral haemorrhage. Cochrane Database Syst Rev. 2023 Jan 26;1(1):CD012144. doi: 10.1002/14651858.CD012144.pub3. PMID 36700520